CLINICAL TRIAL: NCT06294288
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Escalating Single and Multiple Doses of LP-003 in Healthy Volunteers
Brief Title: A Study of Single and Multiple Doses of LP-003 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-10-LP003-2022-01
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: LP-003 Dose 1 (Single) (Experimental)
  Interventions: Biological: LP-003 Dose 1 (Single)
- Cohort 2: LP-003 Dose 2 (Single) (Experimental)
  Interventions: Biological: LP-003 Dose 2 (Single)
- Cohort 3: LP-003 Dose 3 (Single) (Experimental)
  Interventions: Biological: LP-003 Dose 3 (Single)
- Cohort 4: LP-003 Dose 4 (Single) (Experimental)
  Interventions: Biological: LP-003 Dose 4 (Single)
- Cohort 5: LP-003 Dose 5 (Single) (Experimental)
  Interventions: Biological: LP-003 Dose 5 (Single)
- Cohort 6: Placebo (Single) (Placebo Comparator)
  Interventions: Biological: Placebo (Single)
- Cohort 7: LP-003 Dose 6 (Multiple) (Experimental)
  Interventions: Biological: LP-003 Dose 6 (Multiple)
- Cohort 8: LP-003 Dose 7 (Multiple) (Experimental)
  Interventions: Biological: LP-003 Dose 7 (Multiple)
- Cohort 9: LP-003 Dose 8 (Multiple) (Experimental)
  Interventions: Biological: LP-003 Dose 8 (Multiple)
- Cohort 10: Placebo (Multiple) (Placebo Comparator)
  Interventions: Biological: Placebo (Multiple)

INTERVENTIONS:
Biological: LP-003 Dose 1 (Single) — A single dose of LP-003 (Dose 1) was administered intravenously.
  Arms: Cohort 1: LP-003 Dose 1 (Single)
Biological: LP-003 Dose 2 (Single) — A single dose of LP-003 (Dose 2) was administered intravenously.
  Arms: Cohort 2: LP-003 Dose 2 (Single)
Biological: LP-003 Dose 3 (Single) — A single dose of LP-003 (Dose 3) was administered intravenously.
  Arms: Cohort 3: LP-003 Dose 3 (Single)
Biological: LP-003 Dose 4 (Single) — A single dose of LP-003 (Dose 4) was administered intravenously.
  Arms: Cohort 4: LP-003 Dose 4 (Single)
Biological: LP-003 Dose 5 (Single) — A single dose of LP-003 (Dose 5) was administered intravenously.
  Arms: Cohort 5: LP-003 Dose 5 (Single)
Biological: Placebo (Single) — A single dose of placebo was administered intravenously.
  Arms: Cohort 6: Placebo (Single)
Biological: LP-003 Dose 6 (Multiple) — LP-003 (Dose 6) was administered multiple times subcutaneously.
  Arms: Cohort 7: LP-003 Dose 6 (Multiple)
Biological: LP-003 Dose 7 (Multiple) — LP-003 (Dose 7) was administered multiple times subcutaneously.
  Arms: Cohort 8: LP-003 Dose 7 (Multiple)
Biological: LP-003 Dose 8 (Multiple) — LP-003 (Dose 8) was administered multiple times subcutaneously.
  Arms: Cohort 9: LP-003 Dose 8 (Multiple)
Biological: Placebo (Multiple) — Placebo was administered multiple times subcutaneously.
  Arms: Cohort 10: Placebo (Multiple)

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, immunogenicity, pharmacokinetics, pharmacodynamics, and efficacy of LP-003 in healthy volunteers. The study will be conducted in 2 parts: Part 1, the single ascending dose (SAD) is the first in human (FIH) study of LP-003 and Part 2, multiple ascending dose (MAD).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged 18 through 50 years
2. Male subjects must weigh ≥50 kg, and female subjects must weigh ≥45 kg, with a BMI between 19.0 and 28.0 kg/m² (inclusive).
3. Male subjects and their partners or female subjects must agree to use one or more non-pharmaceutical contraceptive methods (such as total abstinence, condoms, Iuds, partner ligation, etc.) during the trial period and for 6 months after the trial, and do not plan to donate sperm or eggs.
4. The subjects fully understand the purpose, nature, method and possible adverse reactions of the experiment, and voluntarily participate in the experiment and sign the informed consent.
5. The subjects were able to communicate well with the researchers and complete the study according to the protocol.

Exclusion Criteria:

1. People who are allergic to the experimental drug and any of its excipients, have a history of allergy to monoclonal antibodies, and are allergic to multiple drugs and food.
2. Patients who have been or are currently suffering from any clinically serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatric and metabolic abnormalities, or any other diseases that can interfere with the test results.
3. Patients who had undergone surgery within 3 months before the trial that the researchers judged would affect drug absorption, distribution, metabolism, and excretion, or had surgery within 4 weeks prior to the trial, or planned to have surgery during the study period.
4. Any history of infection within 14 days prior to administration.
5. A person who is currently infected with parasites or has traveled to an endemic area within the last 3 months or 24 weeks prior to administration.
6. Pregnant and lactating women.
7. Hepatitis B surface antigen, hepatitis C virus antibodies, human immunodeficiency virus antibodies, treponema pallidum antibodies A positive person.
8. Patients who have received any biological agent (including antibodies or derivatives such as omalizumab) within 16 weeks prior to administration (or 5 half-lives, selecting the longer time period).
9. Participants who had participated in other clinical trials within 3 months prior to screening.
10. The investigator deems any condition unsuitable for study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Adverse events | Observation for 280 days after administration
  Number of subjects with treatment-related Treatment Emergent Adverse Events (TEAEs).

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) of LP-003 | Observation for 280 days after administration
  The time when the blood drug concentration reaches its peak after a single dose of medication.
Maximum concentration (Cmax) of LP-003 | Observation for 280 days after administration
  The maximum concentration of LP-003 in the bloodstream after administration.
Elimination half-life (t1/2) of LP-003 | Observation for 280 days after administration
  The time required for the concentration of LP-003 in the bloodstream to decrease by half.
Area under the concentration-time curve (AUC0-t) of LP-003 | Observation for 280 days after administration
  The area under the concentration-time curve (AUC) from time zero to the last chosen time point represents the integral of the drug concentration in the bloodstream over the specified duration.
Apparent clearance rate (CL/F) of LP-003 | Observation for 280 days after administration
  The ratio of drug clearance to drug concentration, represents the apparent clearance of a drug after administration, adjusted for bioavailability.
Assessment of immunogenicity | Observation for 280 days after administration
  The proportion of anti drug antibody (ADA) positive subjects at different detection time points.
Assessment of total immunoglobulin E (IgE) | Observation for 168 days after administration
  The changes in serum total immunoglobulin E (IgE) levels compared to baseline at different assessment time points.
Assessment of free IgE | Observation for 168 days after administration
  The changes in serum free IgE levels compared to baseline at different assessment time points.

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Ding, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No